CLINICAL TRIAL: NCT05863702
Title: Staying Healthy With Follow-up Care: A Feasibility Study Utilizing a Chatbot (Penny) Via Mobile Phones to Increase Compliance With Risk Based Survivorship Care (RBSC) Among Adult Survivors of Pediatric and Young Adult Cancers
Brief Title: Staying Healthy With Follow-up Care: A Mobile Chatbot Feasibility Study for AYA Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UPCC#: 11923
Record Dates: First submitted 2023-04-24; First posted 2023-05-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Survivorship
Keywords: Survivorship; Pediatric Cancers; Young Adult Cancers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention)
- Penny text-messaging program (Experimental)
  Interventions: Behavioral: Penny

INTERVENTIONS:
Behavioral: Penny — The chatbot will assist patients who have not been see for cancer follow-up care, with scheduling follow-up appointments, labs, scans, specialty appointments, and monitor compliance with the appointments made.
  Arms: Penny text-messaging program

SUMMARY:
The purpose of this project is to identify effective strategies to assist survivors of childhood and young adult cancers (diagnosed between birth and age 39) who have not returned for follow-up cancer care for 3 or more years, to reengage with the health care system. The investigator will evaluate the effect of a novel, bidirectional conversational agent ("Penny"), compared to usual care, to assist patients with scheduling appointments, lab work as well as scans and specialty appointments as needed.

DETAILED DESCRIPTION:
To achieve this, the investigator will use a two-arm randomized controlled trial to explore how multilevel factors impact the acceptability and effectiveness of this strategy by collecting qualitative and quantitative data from patients. Penny is a conversational agent ("chatbot") that engages patients in real time via text messaging, allowing for bidirectional communication and motivational cues to promote adherence. The chatbot will assist patients who have not been see for cancer follow-up care, with scheduling follow-up appointments, labs, scans, specialty appointments, and monitor compliance with the appointments made.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age > 18 years), male or female, diagnosed with cancer as a child or as a young adult, between birth and 39 years of age
* Patient possession of a mobile device that can receive SMS texts
* Ability to respond to questions and engage with "Penny" in English
* Ability to provide informed consent to participate in the study
* Approval of the patient's oncology care team for the patient to be involved in the study

Exclusion Criteria:

* Anyone who does not meet the inclusion criteria
* Patients with a history of thyroid cancer or skin cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the utilization of a chatbot (Penny) to increase receipt of evidence-based survivorship care in YA survivors of pediatric and YA cancers | 1 year
  We will identify adult survivors of pediatric and YA cancers who have not been seen for follow-up care >3 years and evaluate patients' engagement with Penny to schedule return appointments and adhere to recommended life-long ongoing follow-up care according to the NCCN guidelines. Patients will be monitored over a 16-week period to see if they scheduled a follow-up care appointment.
Number of patients who agree to use Penny and patient engagement overtime in those patients randomized to the Penny arm | 1 year
  Percentage of initial responses to the conversation initiated by Penny (opt in vs. opt out) providing permission for text messaging
Number of patients who agree to use Penny and patient engagement overtime in those patients randomized to the Penny arm | 1 year
  Total number of times patients engage with Penny to schedule follow up appointments, scans, labs, recommendations for other services made at each clinical visit
Number of patients who agree to use Penny and patient engagement overtime in those patients randomized to the Penny arm | 1 year
  Total number of patients who engage with Penny throughout the study, schedule and are compliant with appointments, scans, labs, and referrals to other services made at each clinical visit

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No